CLINICAL TRIAL: NCT02939833
Title: Effects of Scalp Nerve Blocks on Systemic Inflammation After Meningeoma Resection Surgery：a Prospective Randomized Controlled Trial
Brief Title: Effects of Scalp Nerve Blocks on Systemic Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB20161010
Record Dates: First submitted 2016-10-11; First posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-10

CONDITIONS: Meningiomas
MeSH Terms: conditions — Meningioma | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ropivacaine (Experimental): patients in this group will receive scalp nerve blocks with 0.5% ropivacaine after anesthesia induction and before skull-pin insertion
  Interventions: Procedure: Scalp Nerve Blocks With Ropivacaine
- saline (Placebo Comparator): patients in this group will receive scalp nerve blocks with 0.9% saline after anesthesia induction and before skull-pin insertion
  Interventions: Procedure: Scalp Nerve Blocks With Saline

INTERVENTIONS:
Procedure: Scalp Nerve Blocks With Ropivacaine
  Arms: ropivacaine
Procedure: Scalp Nerve Blocks With Saline
  Arms: saline

SUMMARY:
Patients undergoing meningeoma resection surgery will be randomly assigned to two groups. One group will receive scalp nerve blocks with 0.5% ropivacaine, whereas the other group will receive scalp nerve blocks with 0.9% saline after anesthesia induction and before skull-pin insertion. Serum levels of TNF-α、IL-6 and IL-1β will be measured and compared at before surgery, 1h, 24h and 72h after surgery, respectively. VAS score, dosage of pain-control medicine and NRS score at the first three days after surgery, ratio of intracranial infection within 30d after surgery, and total hospitalization days and medical expenditure will also be recorded and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-28 kg/m2 ASA Physical Status 1-2 diagnosed Meningeoma and will have selective Meningeoma Resection Surgery the incision will be conducted at the frontal, top or the temperal skull.

Exclusion Criteria:

* previous brain surgery severe systemic disease (heart, lung, kidney, or immune system) nerval or mental disorders a history of addiction to opioids allergic to ropivacaine infection at block site or severe systemic infection refuse to attend the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-06 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
serum TNF-α level | 24 hour after surgery
serum IL-6 level | 24 hour after surgery
serum IL-1β level | 24 hour after surgery

SECONDARY OUTCOMES:
serum TNF-α level | 1 hour after surgery
serum IL-6 level | 1 hour after surgery
serum IL-1β level | 1 hour after surgery
serum TNF-α level | 72 hour after surgery
serum IL-6 level | 72 hour after surgery
serum IL-1β level | 72 hour after surgery
VAS score | 24 hour after surgery
VAS score | 48 hour after surgery
VAS score | 72 hour after surgery
dosage of pain-control medicine | within 72 hour after surgery
NRS score | 24 hour after surgery
NRS score | 48 hour after surgery
NRS score | 72 hour after surgery
incidence of intracranial infection | within 30 days after surgery
Hospitalization Days | up to 30 days
out of pocket expenditure for hospitalisation | hospital discharge/up to 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Renji hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided